CLINICAL TRIAL: NCT05185063
Title: Developing a Digital Handover Application for Paramedics to Provide a Personalized Approach to Pre-hospital Stratification for Out of Hospital Cardiac Arrest
Acronym: RAPID-MIRACLE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: London Ambulance Service NHS Trust (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 301864
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Out of Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Out of Hospital Cardiac Arrest
  Interventions: Diagnostic Test: Point of Care blood test

INTERVENTIONS:
Diagnostic Test: Point of Care blood test — The pH will be incorporated into the MIRACLE2 score in a pre-hospital setting. The patients will continue to be treated with standard of care.

SUMMARY:
A prospective study validating the role of the MIRACLE2 score in patients with resuscitated out of hospital cardiac arrest in a pre-hospital setting.

DETAILED DESCRIPTION:
Design: Prospective observational cohort study enrolling OOHCA patients across London in a pre-hospital setting

Study Protocol: Patients with OOHCA and ROSC will be recruited from the community into the study by London Ambulance Service NHS Trust (LAS). LAS has -40 Advanced Paramedic Practitioners in Critical Care (APP-CC) who have a range of specialist skills including airway management and focused ultrasound and attend to over 1500 OOHCAs/year.

Point of Care pH test: The recruited participants will have point of care pH testing performed using the CG4+ iStat system (Abbott Vascular, Illinois, U.S.A.). The test requires 2ml of venous blood and can provide blood results within minutes. The device and blood taking system have received CE marking and are already in routine use across the NHS. Once the blood results are received, the blood sample and testing system are discarded in a routine manner.

Standard Care: Participants will then be conveyed to either the local emergency department or to a HAC based on current routine protocols. Patients will be treated in a routine manner after reaching secondary care in accordance with local and national guidance with no change in care based on this study.

Power calculation: In 2019, APP-CCs from LAS attended to -700 OOHCA patients with ROSC. Assuming 60% recruitment, we could comfortably envisage -500 patients to be recruited in a 15 month period. From previous data, we can expect approximately 60% of the patients (n=300) to have a CPC score of 3-5 on hospital discharge. This would be of a similar size to the dataset used to derive the original score, which gave good levels of accuracy in model performance measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with out of hospital cardiac arrest with sustained ROSC (defined as >20 minutes or sufficient stability to consider conveyance)

Exclusion Criteria:

* Any clear non-cardiac cause of arrest (trauma, drowning Overdose, asphyxia, asthma, anaphylaxis).
* Suspected or confirmed intra-cerebral bleeding
* Known CPC score 3 or 4 pre-cardiac arrest
* Known disease limiting survival to 6 months
* Suspected or known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community (i.e. pre-hospital study)
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral Performance Category at 30 days | 40 dats
  Cerebral Performance Category

SECONDARY OUTCOMES:
All cause mortality at 30 days | 30 days
  Death from any cause
Cause of Death at 30 days | 30 days
  Cause of death defined as neurological,multi-organ dysfunction syndrome, cardiac or unrelated
Cerebral Performance Category at 6 months | 6 months
  Cerebral Performance Category
All cause mortality at 6 months | 6 months
  Death from any cause
Cause of Death at 6 months | 6 months
  Cause of death defined as neurological,multi-organ dysfunction syndrome, cardiac or unrelated

CONTACTS AND LOCATIONS:
Overall Officials: Nilesh Pareek, MA,MRCP,PhD, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Heart Research United Kingdom - Novel Emerging Technology Grant — https://heartresearch.org.uk/improving-care-for-out-of-hospital-cardiac-arrest-oohca-patients-the-rapid-miracle-study/